CLINICAL TRIAL: NCT04970758
Title: Differential Diagnosis Athlete's Heart From Hypertrophic Cardiomyopathy With T1 Mapping
Brief Title: Differential Diagnosis Athlete's Heart From Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019298
Record Dates: First submitted 2021-06-28; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Athlete's Heart

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Athletes /strength exercise
- control group

INTERVENTIONS:
Other:  — no intervention
  Groups: study group

SUMMARY:
Assess the effects of strength sport to heart structure and function by T1 mapping with cardiac resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Same exercise

Exclusion Criteria:

* Intolerance test

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletes
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
T1 value in ms (Unit) | one year
  indicator of the degree of myocardial fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: xinyu wang, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No